CLINICAL TRIAL: NCT05539352
Title: Reducing Suicide Risk in Older Veterans With Mental Health Disorders Using Problem Solving Therapy
Brief Title: Improving Caregivers' Ability to Manage Life Stress
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Supplemental pilot not opened to recruitment due to efforts focusing on primary clinical trial, funding terminated
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MHBC-003-20S-1
Record Dates: First submitted 2022-09-06; First posted 2022-09-14 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Suicidal Ideation
Keywords: caregiver; Cognitive Behavioral Therapy; suicidal ideation; suicide prevention; executive functioning; functional disability
MeSH Terms: conditions — Suicidal Ideation; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: The study design is a single arm, receiving PST+EUC. Both parts of the treatment are evidence-based interventions, and the treatment protocol is delivered in six sessions. The study will occur at VA Palo Alto.
Masking Description: This is a single-arm pilot study with no random assignment to groups. No masking is applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active treatment plus EUC (Experimental): All caregivers are assigned to this condition and receive the treatment plus EUC.
  Interventions: Behavioral: Problem Solving Therapy (PST) plus EUC

INTERVENTIONS:
Behavioral: Problem Solving Therapy (PST) plus EUC — All caregivers are assigned to this condition and receive EUC and PST. EUC is delivered along with the treatment to ensure the safety of all caregivers enrolled in the study. In addition to EUC, caregivers receive PST, which teaches patients a structured "planful problem solving" approach to: 1) identify problems and set goals, 2) generate alternative solutions, 3) select a solution based on cost-benefit analysis, and 4) devise and implement a plan for the solution and assess its effectiveness in solving the problem. This contemporary PST protocol also teaches tool kits to address obstacles highly pertinent to the challenges faced by caregivers and active suicidal ideation: emotion dysregulation, hopelessness, and feeling overwhelmed by too much information ("brain overload") or stress.
  Other Names: PST plus EUC

SUMMARY:
The COVID-19 pandemic has led to increased caregiving demands for caregivers of Veterans with dementia. Dementia caregivers are particularly at-risk for depression and anxiety, known risk factors for increased suicidality. Emerging research also suggests that dementia caregivers are experiencing greater suicidality during COVID-19 at a time when VHA is also devoting increased efforts toward caregiver health and support services. Aims are to determine the feasibility and acceptability of video-delivered Problem-Solving Therapy for reducing suicide risk in caregivers of Veterans with dementia.

DETAILED DESCRIPTION:
The proposed single-arm pilot will examine the feasibility and acceptability of a brief behavioral treatment for reducing suicidal ideation and for increasing reasons for living in caregivers of Veterans with dementia. The proposed study will examine Problem Solving Therapy (PST) using a protocol that teaches skills to address emotional and practical barriers to effective problem solving. The VA usual care practice of collaborative safety planning will also be included in the treatment protocol, herein referred to as enhanced usual care (EUC). For participant safety, all caregivers will receive both PST and EUC. The study design is a single arm. Both PST and EUC are evidence-based interventions, and the treatment is delivered in six sessions. The study will occur at VA Palo Alto.

The assessments and treatments will be conducted entirely by video. Participants will be sent VA-approved tablets. Longitudinal assessment of suicidal ideation and reasons for living will occur at eleven timepoints: baseline, after each of the six weekly treatment sessions, posttreatment (7 weeks), at 1-, 3-, and 6-month follow-up. The recruitment goal is 10 caregivers. Caregivers must be 50 years or older and report suicide ideation to be eligible. Veterans will be excluded and referred for other services if they have psychotic symptoms, bipolar disorder, or severe OCD; an alcohol/substance use disorder; severe or unstable medical conditions; recent head injury (past year) or history of a head injury with loss of consciousness for 24 or more hours; terminal illness; positive cognitive screen indicative of possible dementia; or if they are unable to participate in the study or follow-up sessions. Recruitment will occur through multiple strategies at VA, Vet centers, and in the community to ensure the feasibility of recruiting a total of 10 caregivers.

ELIGIBILITY:
Inclusion Criteria:

* 50 years old or older
* Identify as a informal caregiver to at least 1 older Veteran
* SI (past month) on the C-SSRS. No SI or imminent risk (will be excluded). Eligibility includes non-specific active suicidal thoughts to active SI with some planning (on C-SSRS item 3: "Have you been thinking about how you might do this") and/or some intent to act (on C-SSRS item 4: "Have you had these thoughts and had some intention of acting on them?") provided that those endorsing item 4 have an established relationship with a psychiatrist aware of this intent level (who is not also performing psychotherapy). Those endorsing C-SSRS item 5: "Do you intend to carry out this plan?" would be considered at imminent risk and excluded. No suicide attempt in the past 3 months.
* No diagnosis of dementia; evidence that cognitive impairment is not indicative of possible dementia based on a negative cognitive telephone screen (<10 errors on the Blessed cognitive screen)
* No diagnosis on MINI or medical record for psychotic symptoms or disorders, bipolar disorder, or severe OCD (mild or moderate OCD will be eligible).
* No history of head injury past 12 months or no lifetime history of head injury with LOC > 24 hours
* No severe or unstable chronic medical illness or other severe or unstable respiratory, cardiovascular, neurologic, hepatic, hematopoietic, gastrointestinal or metabolic dysfunction
* AUDIT Total cut-off scores for inclusion of 14 or lower for men, and 12 or lower for women (no current alcohol use disorder)
* No prominent homicidal ideation
* English language proficiency to engage in treatment
* Sensory abilities sufficiently intact to engage in assessment and treatment
* Not currently enrolled in psychotherapy for a mental health issue (see details below in Exclusion Criteria)
* No current prescription for anti-psychotics if prescribed for a psychotic disorder. Anti-psychotics for depression without psychosis are eligible. Psychotropic medications (e.g., SSRIs) are also eligible. Medication changes are allowed after study enrollment
* Participants must not meet criteria for any substance use disorder for illicit substances, as determined by the MINI. Further, participants must not meet criteria for moderate or severe substance use disorder for cannabis/marijuana (mild substance use disorder may be included)

  * Access to internet connection in a private area (e.g., own or other's home, office, etc.) to engage in private online treatment sessions by video. Does not need video/internet-enabled device (study will provide a tablet), just access to internet

Exclusion Criteria:

* Less than 50 years old
* No SI (past month) or imminent risk on the C-SSRS will be excluded. Those endorsing C-SSRS item 5: "Do you intend to carry out this plan?" would be considered at imminent risk and excluded. Exclude if there is a suicide attempt in the past 3 months
* Diagnosis of dementia; evidence that cognitive impairment is indicative of possible dementia based on a positive cognitive telephone screen (>=10 errors on the Blessed cognitive screen)
* Diagnosis on MINI or medical record for psychotic symptoms or disorders, bipolar disorder, or severe OCD (mild or moderate OCD will be eligible).
* History of head injury past 12 months or lifetime history of head injury with LOC > 24 hours
* Severe or unstable chronic medical illness or other severe or unstable respiratory, cardiovascular, neurologic, hepatic, hematopoietic, gastrointestinal or metabolic dysfunction
* AUDIT Total cut-off scores for exclusion to scores of 15 or higher for men, and 13 or higher for women (no current alcohol use disorder)
* Prominent homicidal ideation
* Lacking English language proficiency to engage in treatment
* Sensory abilities not sufficiently intact to engage in assessment and treatment
* Currently enrolled in psychotherapy for a mental health issue: Participants will be excluded if they are currently enrolled in some other individual psychotherapy or evidence-based group therapy (e.g., cognitive behavioral therapy for depression), but the participant would be eligible for the study after they complete their treatment if they still have suicidal ideation. Participants who are receiving mental health care are eligible if their current care includes treatment from a psychiatrist, supportive therapy, peer counseling or support, or participating in psychoeducational groups. Once enrolled in the study, unless there is an unanticipated contraindication to continue the participant in the study while they are receiving other mental health care, they will be retained in the study. Participants will stop study treatment if there is any contraindication to continue the participant in the study while they are receiving new mental health treatment outside of the study.
* Current prescription for anti-psychotics
* Individuals who meet criteria for any substance use disorder for illicit substances or for moderate or severe substance use disorder for cannabis/marijuana will be excluded

  * Lack of access to internet connection in a private area (e.g., own or other's home, office, etc.); inability to engage in private online treatment sessions by video

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment and retention of participants | At study completion, up to 41 months or completed participation of all participants, whichever came first
  The investigators will estimate the rate of recruitment during the course of the study, to inform feasible recruitment rates for future clinical trials with this population. Feasibility of retention will be established if 80% or more of enrolled participants are retained for at least 5 of 6 treatment sessions.
Appropriateness of inclusion/exclusion criteria | At study completion, up to 41 months or completed participation of all participants, whichever came first
  Appropriateness of the inclusion/exclusion criteria will be determined by examining frequency tables and/or qualitative data indicating number and types of reasons for screening failures and withdrawals from the treatment/study. These frequency tables will inform decisions in future research regarding modifications to inclusion/exclusion criteria.
Acceptability of treatment | At posttreatment (7 weeks)
  Acceptability of the treatment will be determined based on adherence in attending sessions and completing homework, and treatment satisfaction ratings. A threshold of 80% or more (5 out of 6 sessions attended; 4 or more with completed homework [no homework in first session]), based on the rates reported for other late-life behavioral intervention studies, will be used to establish adherence. Mean ratings of 3 ("good/helpful") or higher on a 5-point item assessing how effective the treatment was in helping participants to deal better with their problems, and mean ratings of 3 ("somewhat met my expectations") or higher on a 4-point item assessing how well the treatment met their expectations, will be used to establish treatment satisfaction. Treatment expectations, likes, and dislikes will be analyzed by identifying themes of patient responses and tallying them in a frequency table for review. This will help determine if certain aspects of the treatments should be retained or modified.

SECONDARY OUTCOMES:
Sensitivity of trial outcome measures | Change from baseline to posttreatment (7 weeks)
  Sensitivity of the potential outcome measures for future randomized clinical trials will be determined. Mean pre- and post-scores will be compared using t-tests to determine the direction of change on the following measures: Geriatric Suicide Ideation Scale (GSIS), Reasons for Living - Older Adults Scale (Short RFL-OA), WHO Disability Assessment Schedule (WHO-DAS 2.0) short form, DKEFS Verbal Fluency Test, WAIS Digit Span subtest (Digits Forward and Backward), Oral Trail Making Test.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A Beaudreau, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. The data set will be shared upon written request and will be shared pursuant to a Data Use Agreement (DUA) once the planned manuscripts have been accepted to peer-reviewed journals. At that time, the investigators will send researchers who have completed a DUA a electronic copy of the database in a password protected database file. Final datasets will be maintained locally until VA enterprise-level resources become available for long term storage and usage.
Supporting Information: Study Protocol, ICF
Time Frame: Publications from this project will be made available through the National library of Medicine PubMed Central website 1 year of the date of publication. The final de-identified datasets underlying these publications will be available by written request to the PD/PI. Data will be available by written request until March 31, 2046. This date will be extended if it is determined that availability of the data to researchers would be in the interest of the scientific literature on suicide prevention, or if additional research questions can be developed the data to address important gaps in suicide prevention assessment and treatment.
Access Criteria: Protection of privacy, confidentiality, and proprietary data is ensured using the following mechanisms: 1) a de-identified dataset, 2) signed data user agreement that will prohibit researchers requesting the data from identifying or attempting to re-identify individuals in the dataset ,3) "90+" age category, but not an exact age for adults aged 90 years or older to prevent identification, 4) sharing only of quantitative data, but not qualitative data to further prevent identification.